CLINICAL TRIAL: NCT06081751
Title: The Effect of Traditional Children's Games on Internet Usage Time and Stress Level of Primary School Students; Randomized Controlled Study
Brief Title: The Effect of Traditional Children's Games on Internet Use Stress Level of Primary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serap Batı, Dr. Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sbati
Record Dates: First submitted 2023-08-28; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Internet; Stress Level
Keywords: stress; internet; traditional children's games
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Children in the intervention group will play traditional games for 60 minutes, 3 days a week for 8 weeks. The program to be implemented is as follows;
  Week 1 (Day 1 - I Sell Oil, I Sell Honey game, Day 2 - Snatch game, Day 3 - Corner Snatch Game) Week 2 (Day 1 - Handkerchief game, Day 2 - My Fire game, 3 Day 2 - Kurt Baba Game) Week 3 (Day 1 - Chubby game, Day 2 - Jump rope game, Day 3 - Mouse game in the middle) Week 4 (Day 1 - Rook dodgeball game, Day 2 - Stop game, Day 3 - Old cushion mouse game) Week 5 (Day 1 - I Sell Oil, I Sell Honey game, Day 2 - Snatch game, Day 3 - Corner Catch Game) Week 6 (Day 1 - Handkerchief grabbing game, Day 2 - My Fire game, Day 3 - Daddy Wolf Game) Week 7 (Day 1 - Chubby game, Day 2 - Jumping rope game, Day 3 - Mouse game in the middle) Week 8 ( Day 1 - Dodgeball game, Day 2 - Stopping game, Day 3 - Old matte mouse game)
  Interventions: Behavioral: Pretest; Behavioral: Posttest
- Control Group (Active Comparator): no intervention will be made
  Interventions: Behavioral: Pretest; Behavioral: Posttest

INTERVENTIONS:
Behavioral: Pretest — Internet usage time, "How many hours do you use the Internet per day?" and "What is your weekly internet usage frequency?" will be questioned using questions.
  Child Perceived Stress Scale was developed by Snoeren-Hoefnagels (2014) and adapted to Turkish by Oral and Ersan in 2017. The scale consists of 9 items. It is a 4-point Likert type scale. It consists of a single sub-dimension. The answer "never" gets one point, and the answer "always" gets 4 points. In the scale that does not contain reverse items, the minimum score is 9 and the maximum score is 36. High scores from the scale questions mean that the individual's stress level is high.
  I
  Other Names: Questionnaire (Including Internet Usage Time,Child Perceived Stress Scale )
Behavioral: Posttest — Internet usage time, "How many hours do you use the Internet per day?" and "What is your weekly internet usage frequency?" will be questioned using questions.
  Child Perceived Stress Scale was developed by Snoeren-Hoefnagels (2014) and adapted to Turkish by Oral and Ersan in 2017. The scale consists of 9 items. It is a 4-point Likert type scale. It consists of a single sub-dimension. The answer "never" gets one point, and the answer "always" gets 4 points. In the scale that does not contain reverse items, the minimum score is 9 and the maximum score is 36. High scores from the scale questions mean that the individual's stress level is high.
  I
  Other Names: Questionnaire (Including Internet Usage Time, Child Perceived Stress Scale)

SUMMARY:
Traditional games are games based on interpersonal communication and creativity, mostly involving physical activity. These aspects have positive contributions to the development of the child. Studies show that group games that include physical activity cause a decrease in children's stress levels. Playing as a team member and working for a common goal can contribute to the social development of the child.

Today, with the development of technology, the interest in games played with the internet has increased, which has caused children to be drawn from the streets to their homes. Turning to internet games also prevents children from socializing and causes them to lead a sedentary life. Spending more time on internet games causes sleep problems, conflict with family members, decrease in school success, increase in stress level, and delay in social skills. It is stated that nurses have important responsibilities in preventing excessive internet use, which affects children's physical, mental and social development. It is thought that this study will help children spend their free time with activities that will positively affect their development through traditional children's games, and thus contribute to the reduction in internet usage times and stress levels.

DETAILED DESCRIPTION:
Today, with the development of technology, the interest in games played with the internet has increased, which has caused children to be drawn from the streets to their homes. Turning to internet games also prevents children from socializing and causes them to lead a sedentary life. Spending more time on internet games causes sleep problems, conflict with family members, decrease in school success, increase in stress level, and delay in social skill. It is stated that nurses have important responsibilities in preventing excessive internet use, which affects children's physical, mental and social development. It is thought that this study will help children spend their free time with activities that will positively affect their development through traditional children's games, and thus contribute to the reduction in internet usage times and stress levels.

MATERIALS AND METHODS Purpose of the research The research was carried out to determine the effect of traditional children's games on internet usage time and stress level.

hypotheses H0 a = There is no difference in the duration of internet use between the experimental and control groups.

H0 b = There is no difference between the total scores of the Perceived Stress Scale in Children (8-11 years) between the experimental and control groups.

Type of Research The research is a pre-test, post-test, parallel group, randomized controlled study to determine the effect of traditional children's games on internet usage time and stress level.

Location and Characteristics of the Research The research was carried out in Seydişehir Mahmut Esat Secondary School affiliated to Konya Provincial Directorate of National Education. The reason for choosing this school is that it is one of the schools with a high number of students in the district of Seydişehir and has easy transportation. There are 1079 students enrolled in Seydişehir Mahmut Esat Secondary School in the 2021-2022 academic year. The school has a total of 18 classes and 516 students, nine of which are in the 5th and 6th grades, and nine are in the 6th grade. Schools provide full-time education. There are no infirmaries and nurses in schools. School gardens and gymnasiums are adequate for play.

Population and Sample of the Research The universe of the research consisted of 516 students enrolled in the 5th and 6th grades in the related school in the 2022-2023 academic year. The reason for the inclusion of students in this age group in the study is that they use the game as a tool to reflect the developmental characteristics of the children. For the study group of the experimental research, a computer-assisted simple random numbers table was prepared by an independent statistics expert among 516 students. 108 students were selected by simple random sampling. 30 students included in the study were randomly assigned to the experimental and 30 control groups.

The work will be carried out in two stages. In the first stage, Parental Consent Form", "Descriptive Characteristics Form" will be sent to the families of the students at the school. According to the answers from the parents, the children's internet usage time and frequency will be determined, and students with more internet usage time (more than 2 hours a day) and frequency (who use the internet every day) will be included in the sample.

The sample size of the study was calculated based on the results of different studies:

In a study examining the effects of traditional children's games on internet addiction, social skills and stress levels, the stress post-test mean scores of the group that played and did not play traditional games were 75±43.15 in the experimental group and 253.31±29.19 in the control group. According to these values, it was calculated that the sample size should be at least 60 (30/30) with an effect size of 0.77, a power of 0.80 and a margin of error of 0.05, according to the calculation made in the G*Power 3.1.4 package program.

Randomization After obtaining their consent and pre-testing, the 60 students who make up the study group of the experimental research will create a random number sequence by an independent statistician and will be assigned to the experimental (30) and control (30) groups with a simple randomization method (www.randomizer.org). A separate randomization table for girls and boys was created from the created class list (Table 4).

CONSORT CHART This study is a randomized controlled pretest-posttest study. It has been planned in accordance with the CONSORT criteria.

Inclusion Criteria for Participants in the Study

* Approval by the student's family to participate in the study
* Internet usage time is more than 2 hours a day and its frequency is every day
* Willingness to participate in the research Criteria for Exclusion of Participants in the Study
* Having a physical, orthopedic or mental illness or disability that may interfere with playing
* Regularly participating in sporting events
* Occurrence of unwanted injury during traditional children's games
* Not being able to attend the traditional children's play program for at least two weeks.

Data Collection Technique and Tools In the collection of research data; The descriptive features form developed by the researchers and the perceived stress scale in children (8-11 years) will be used.

Descriptive Characteristics Form It includes socio-demographic information about the child and parent, and information about the duration of internet use.

Perceived Stress Scale in Children (8-11 years) It was developed by Snoeren-Hoefnagels (2014) and adapted into Turkish by Oral and Ersan in 2017. When the child evaluates the past week, he is asked to give answers about how appropriate each item is for him. The scale consists of 9 items. It is a 4-point Likert scale. It consists of a single sub-dimension. Responses to the items were graded as 'never', 'sometimes', 'often' and 'always'. Never gets one point and always gets 4 points. A minimum score of 9 and a maximum score of 36 are obtained in the scale without reversed items. High scores on the scale questions mean that the individual's stress level is high.

Data Collection Data Collection Pre-tests will be applied after obtaining written consent from the experimental and control groups in the 2022-2023 academic year. After the application program is completed, the final tests will be applied to the experimental and control groups.

Application of Research Experimental group The study will be carried out in the 2021-2022 academic year after the necessary permissions are obtained. Before the application, information will be given by meeting with the school administration and teachers. In a closed envelope to the parents of the students in the intervention and control groups;

* Parental Consent Form
* A Descriptive Characteristics Form will be sent and parents who agree to participate in the study will be asked to fill in the other forms in the envelope. The envelopes sent will be collected by the teachers after 1 week.

Students who were allowed to participate in the study with a consent form by their parents and who have more internet usage time (more than 2 hours a day) and frequency (who use the internet every day) according to the data specified in the "Descriptive Characteristics Form" will be included in the study. The "Perceived Stress Scale for Children (8-11 Years)" will be administered to the children included in the sample.

Children in the intervention group will be played for 60 minutes, 3 days a week for 8 weeks, according to the rules set in the "Traditional Children's Games Festival Games Guide Booklet" prepared by the Ministry of National Education and the Ministry of Youth and Sports.

After the program is completed, the "Perceived Stress Scale for Children (8-11 Years)" will be re-applied to the students, the parents will be sent the Descriptive Characteristics Form again in a closed envelope and asked to fill in, and it will be collected by the teachers 1 week later.

No attempt will be made on the control group. Pre-test-post-tests will be applied in parallel with the intervention group at the same time.

blinding Subjects will not be blinded due to the active role of the intervention group in the study. Blinding will be done in statistics and reporting in the research. The input of the research data (pre-tests and post-tests and transferring the data to the computer) will be entered with "A" and "B" codes without specifying the experimental or control group. The analysis of the data will be done by an independent statistician. After the statistical analysis is made and the research report is written, the coding for the experimental and control groups will be explained to the expert by the coder. Researchers will be blinded to statistical analysis until the study is complete.

Variables of the Study Dependent variables: Internet use and stress level Independent variables: Playing traditional children's games Ethical Dimension of Research

* Permission will be obtained from the Ethics Committee of the Faculty of Health Sciences of Necmettin Erbakan University.
* Permission was obtained from the Ministry of National Education.
* Written permission was obtained from the authors for the use of scales.
* Written consent will be obtained from the children's parents.
* Verbal consent will be obtained from children. Limitations of the Research The findings of the study can only be generalized to the universe in which the study was conducted. In the implementation process of the research, there may be difficulties in ensuring the voluntary basis, since the application will be made to the participants during extracurricular times and after school.

Statistical Evaluation of Data The data obtained from the research will be evaluated with the SPSS 20.0 (Statistical Package for Social Sciences) package program. Number, percentage, mean and standard deviation will be used as descriptive statistics in the evaluation of the data. Chi-square test or McNemar test will be used to compare categorical data. In the analysis of the data, Mann Whitney U test will be used in independent groups and Wilcoxon Signed Rank Test will be used in dependent groups. Significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* • Approval by the student's family to participate in the study

  * Completing the Internet Addiction Scale by their families
  * Internet usage time is more than 2 hours a day and its frequency is every day
  * Volunteering to participate in research

Exclusion Criteria:

* • Having a physical, orthopedic or mental illness or disability that may interfere with playing

  * Regular participation in sporting events
  * Occurrence of unwanted injury during traditional children's games
  * Not participating in the traditional children's play program for at least two weeks.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
It is expected that there will be changes in the daily internet usage times of the students in the experimental group. | 8 weeks
  with the survey
It is expected that there will be a change in the "Perceived Stress Scale for Children (8-11 years)" scores of the students in the experimental group. | 8 weeks
  with the survey

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No